CLINICAL TRIAL: NCT07398885
Title: Assessing the Impact of Herbal Supplement on Fatigue and Disease Activity in SLE: Results From an 8-Week Randomized Trial
Acronym: TIR-CUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Tayssir Ben Achour, principal investigator, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTelmanar
Record Dates: First submitted 2024-03-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: System; Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus , Fatigue, EVACUR, Herbal supplement, FACIT-F, SLEDAI, Randomized controlled trial.
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized double-blind clinical trial conducted at various internal medicine services in Tunisia over a period of 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A two -to-one (2:1) randomization was performed in this study in which patients were randomly assigned into two groups: Group 1 (G1) which received EVACUR, and Group 2 (G2) received a placebo. Randomization was handled by an independent third party using a dedicated randomization software.
  Double-Blind Design:
  Neither the patients nor the investigators knew the treatment assignment. EVACUR and placebo capsules are identical in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVACUR (Experimental): EVACUR and the placebo are produced by the Wellnet laboratory. It is a herbal therapy in capsule form. It is a bottle containing 40 capsules composed of: black seed, zinc sulfate, Echinacea, vitamin C, red ginseng, ginger, chamomile, spirulina, royal jelly, Ganoderma, vitamin B1, B6, B12, selenium.
  Ingredient Latin/INCI Name Form/Quality Quantity per capsule Black seed Nigella sativa Dry extract 80 mg Echinacea Echinacea spp. Dry extract 40 mg Ginger Zingiber officinale Dry extract 30 mg Chamomile Matricaria chamomilla Dry extract 10 mg Red ginseng Panax ginseng Dry extract 10 mg Reishi mushroom Ganoderma lucidum Dry extract 10 mg Spirulina Spirulina spp. Dry extract 60 mg Royal jelly Royal jelly Lyophilized 20 mg Vitamin C Ascorbic acid - 30 mg Zinc Zinc sulfate - 2.5 mg Vitamin B1 Thiamine - 3 mg Vitamin B6 Pyridoxine Marine source 4 mg Vitamin B12 Cobalamin - 10 µg Selenium Selenium yeast - 40 µg
  Interventions: Dietary Supplement: EVACUR
- PLACEBO (Placebo Comparator): consists of starch capsules arranged in a bottle that looks identical to that of EVACUR.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: EVACUR — It is a herbal therapy in capsule form. It is a bottle containing 40 capsules composed of: black seed, zinc sulfate, Echinacea, vitamin C, red ginseng, ginger, chamomile, spirulina, royal jelly, Ganoderma, vitamin B1, B6, B12, selenium.
  EVACUR is adminstrated at a rate of 2 capsules per day in the morning
  Arms: EVACUR
Other: PLACEBO — starch capsules arranged in a bottle that looks identical to that of EVACUR. It is administered at a rate of 2 capsules per day in the morning.
  Arms: PLACEBO

SUMMARY:
Fatigue is one of the most prevalent and disabling manifestations of systemic lupus erythematosus. Although its management often entails a combination of pharmacologic and non-pharmacologic strategies, no pharmacologic intervention has yet demonstrated consistent efficacy.

Aim: The purpose of this clinical study was to explore the efficacy of using herbal-based treatment on patients with SLE-related fatigue .

Methods: We performed a 8-week,randomized, double-blinded, placebo-controlled clinical trial in two internal medicine departments in Tunisia over a period of 2 months. We included patients with SLE who met the classification criteria of the 2019-EULAR/ACR classification criteria for SLE and had a FACIT-F (Functional Assessment of Chronic Illness Therapy-fatigue) score minor than 34. After screening, patients were randomly assigned to the EVACUR treatment group or placebo group. The primary endpoints were changes in fatigue (FACIT-F) and disease activity (SLEDAI) scores.

DETAILED DESCRIPTION:
Study Type:

This was a randomized, double-blind clinical trial conducted in two internal medicine departments in Tunisia over a period of 3 months.

Study Population:

Patients with a diagnosis of SLE who were being followed in the participating departments.

Inclusion Criteria:

Age superior than 18 years Confirmed diagnosis of SLE according to the 2019 ACR/EULAR classification criteria Presence of fatigue, defined as a FACIT-F score < 34 Signed informed consent

Non-Inclusion Criteria:

Pregnancy or breastfeeding Diseases or comorbidities that may influence fatigue:untreated hypothyroidism, psychosis common infections, and other autoimmune and inflammatory diseases Patients on vitamin K antagonist therapy, due to a possible interaction with Ginger and Nigella History of severe allergy or intolerance to EVACUR or any component of the placebo

Exclusion Criteria:

Diagnosis of another systemic disease during the study period Pregnancy Allergy to any component of EVACUR Withdrawal of consent

Data Collection:

Patient data were collected from medical records,including epidemiological characteristics such as age at inclusion , gender and medical and family history .Disease-specific data included the duration disease, systemic manifestations,nature of treatement at inclusion .Disease activity was evaluated using clinical SLEDAI-2K score. Baseline FACIT score was collected.Biological assessments were performed such us Anti-dsDNA antibody titers ,ANA and serum C3 and C4 levels.

Study protocol:

Randomization:

A two -to-one (2:1) randomization was performed in this study in which patients were randomly assigned into two groups: Group 1 (G1) which received EVACUR, and Group 2 (G2) received a placebo. Randomization was handled by an independent third party using a dedicated randomization software.

Double-Blind Design:

Neither the patients nor the investigators knew the treatment assignment. EVACUR and placebo capsules are identical in appearance.

Treatement:

EVACUR:

A phytotherapeutic compound presented in capsule form. Each bottle contains 40 capsules composed of: Nigella seed, Zinc sulfate, Echinacea, Vitamin C, Red ginseng, Ginger, Chamomile, Spirulina, Royal jelly, Ganoderma, Vitamins B1, B6, B12, Selenium(Table1).

Contra-indications: Allergy to any component of the supplement. Table 1. Ingredients and Dosage of EVACUR Formulation per Capsule Ingredient Latin/INCI Name Form/Quality Quantity per capsule Black seed Nigella sativa Dry extract 80 mg Echinacea Echinacea spp. Dry extract 40 mg Ginger Zingiber officinale Dry extract 30 mg Chamomile Matricaria chamomilla Dry extract 10 mg Red ginseng Panax ginseng Dry extract 10 mg Reishi mushroom Ganoderma lucidum Dry extract 10 mg Spirulina Spirulina spp. Dry extract 60 mg Royal jelly Royal jelly Lyophilized 20 mg Vitamin C Ascorbic acid - 30 mg Zinc Zinc sulfate - 2.5 mg Vitamin B1 Thiamine - 3 mg Vitamin B6 Pyridoxine Marine source 4 mg Vitamin B12 Cobalamin - 10 µg Selenium Selenium yeast - 40 µg

Placebo:

Capsules containing starch, packaged identically to EVACUR bottles. Both treatments will be administered at a dose of 2 capsules per day in the morning (3 bottles per patient for the study duration).

Follow-up:

Patients attended three visits at baselineM0, one monthM1, and two monthsM2. The FACIT score was assessed during each visit along with a physical examination.

Adverse Events:

Potential side effects will be recorded and evaluated throughout the study. Occurrence of any adverse event will lead to patient exclusion and trigger a pharmacovigilance investigation. All adverse events must be reported immediately to the principal investigator.

Fatigue Assessment Score:

Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) A 13-item questionnaire with responses on a Likert scale from 1 (not at all) to 5 (very much).

Total score out of 52; higher scores indicate less fatigue.Can be calculated if at least 50% of the questions are answered.

Reliability: High (Cronbach's alpha = 0.94) Validity: Strong, with good correlation with other fatigue measurement tools Completion time: 5-10 minutes A validated Arabic version is available with good psychometric properties .

Evaluation Criteria:

Primary Endpoint:

A mean Facit-F score improvement between G1 and G2 at month2 > Minimal Clinically Important Difference(MCID).The MCID in SLE is estimated at 3.4T[5].

Secondary Endpoints:

Improvement in the disease activity SLEDAI score Good tolerance of the dietary supplement.

Statistical Analysis:

Data were analyzed using SPSS.Appropriate statistical tests will be applied, including Student's t-test or the Wilcoxon test.Randomization will be conducted using dedicated software.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed diagnosis of SLE according to the 2019 ACR/EULAR classification criteria
* Presence of fatigue, defined as a FACIT-F score < 34
* Signed informed consent

Non-Inclusion Criteria:

* Pregnancy or breastfeeding
* Diseases or comorbidities that may influence fatigue:untreated hypothyroidism, psychosis common infections, and other autoimmune and inflammatory diseases
* Patients on vitamin K antagonist therapy, due to a possible interaction with Ginger and Nigella
* History of severe allergy or intolerance to EVACUR or any component of the placebo

Exclusion Criteria:

* Diagnosis of another systemic disease during the study period
* Pregnancy
* Allergy to any component of EVACUR
* Withdrawal of consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Tirderness Score: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | at inclusion, after 1, 2 months
  * This is a 13-question questionnaire to which the patient responds on a Likert scale ranging from 1 to 5 (1 = completely, 5 = not at all). By adding up the responses, a score out of 65 is obtained. The higher the score, the less fatigued the patient is [2].
  * The score can be calculated once the patient has answered 50% of the questions.
  * Reliability: The Cronbach's alpha is good (0.94).
  * Validity: This tool has good validity as it has a strong correlation with the use of other scales.
  * It takes 5 to 10 minutes to complete the questionnaire and calculate the score.
  * The Arabic version (Appendix 3) has been validated with good psychometric properties

CONTACTS AND LOCATIONS:
Locations (1):
- La Rabta Hospital, Ben Arous, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cella D, Yount S, Sorensen M, Chartash E, Sengupta N, Grober J. Validation of the Functional Assessment of Chronic Illness Therapy Fatigue Scale relative to other instrumentation in patients with rheumatoid arthritis. J Rheumatol. 2005 May;32(5):811-9. PMID 15868614
- [Background] Al Maqbali M, Hughes C, Gracey J, Rankin J, Hacker E, Dunwoody L. Psychometric Properties of the Arabic Version of the Functional Assessment of Chronic Illnesses Therapy-Fatigue in Arabic Cancer Patients. J Pain Symptom Manage. 2020 Jan;59(1):130-138.e2. doi: 10.1016/j.jpainsymman.2019.10.008. Epub 2019 Oct 21. PMID 31647976
- [Result] Dey M, Parodis I, Nikiphorou E. Fatigue in Systemic Lupus Erythematosus and Rheumatoid Arthritis: A Comparison of Mechanisms, Measures and Management. J Clin Med. 2021 Aug 13;10(16):3566. doi: 10.3390/jcm10163566. PMID 34441861
- [Result] Mertz P, Schlencker A, Schneider M, Gavand PE, Martin T, Arnaud L. Towards a practical management of fatigue in systemic lupus erythematosus. Lupus Sci Med. 2020 Nov;7(1):e000441. doi: 10.1136/lupus-2020-000441. PMID 33214160

DOCUMENTS (1):
  • Study Protocol (2026-01-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT07398885/Prot_000.pdf